Rev: A 

# DS Biopharma Protocol #: DS107G-03

A Randomised, Double-blind, Placebo-Controlled, Phase 2b Study to Assess the Efficacy and Safety of Orally Administrated DS107 in Patients with Moderate to Severe Atopic Dermatitis

# Statistical Analysis Plan

Created by: Clinical Trial Data Services, LLC

40 Nagog Park, Suite #210

Acton, MA 01720

Lavin Consulting LLC 3 Cahill Park Drive Framingham MA 01702



Statistical Analysis Plan DS Biopharma DS107G-03

Rev: A 

By signing the following, I agree to the contents in the Statistical Analysis Plan and its associated attachments.

### Approved by:

| Name | Title | Signature | Date |
|---|---|---|---|
| Phil Lavin, PhD | Senior Biostatistical<br>Consultant (for sponsor) | Philip lan- | 7/17/2017 |
| Terri Sampo, MPH | Principal Consultant,<br>CTDS | Thego | 07/17/2017 |



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

#### LIST OF ABBREVIATIONS

15-HETrE 15-hydroxyeicosatrienoic acid

AD Atopic Dermatitis AE Adverse Event

BD Bis Die (Twice daily)
BD Blood Pressure

BP Blood Pressure
BPM Beats Per Minute

CM Concomitant Medication

COX Cyclooxygenase

CRA Clinical Research Associate
CRO Contract Research Organisation

CRF Case Report Form Cyclosporin A

CDISC Clinical Data Interchange Standards Consortium

CTA Clinical Trial Agreement

DGLA Dihomo-Gamma-Linolenic Acid DLQI Dermatology Life Quality Index

DM Data Manager
DS DS Biopharma

EASI Eczema Area and Severity Index

EC Ethics Committee
EDC Electronic Data Capture
FAS Full Analysis Set

FSH Follicule Stimulating Hormone

GCP Good Clinical Practice

GENMOD Generalized Linear Model (binary outcomes)

GLP Good Laboratory Practice ICF Informed Consent Form

ICH International Conference on Harmonisation

IGA Investigator's Global Assessment

IgE Imunnoglobulin E

IMP Investigational Medicinal Product

ISF Investigator Site File ITT Intention-To-Treat

IWRS Interactive Web Response System MCAR Missing Completely at Random

MedDRA Medical Dictionary for Regulatory Activities
MMRM Mixed Model with Repeated Measures

MNAR Missing Not at Random

NOAEL No Observed Adverse Event Limit

NRS Numeric Rating Scale OTC Over The Counter



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

PBIR Probability of Being in Response

PGD1 Prostaglandin D1

PGI-C Patient Global Impression of Change PGI-S Patient Global Impression of Severity

PIS Patient Information Sheet

PK Pharmacokinetics

POEM Patient Orientated Eczema Measure

PPS Per Protocol Analysis Set PUVA Psoralen & Ultraviolet A

PV CRO Pharmacovigilance Contract Research Organisation

SAE Serious Adverse Event
SAS Statistical Analysis System
SAP Statistical Analysis Plan

SCORAD SCORing AD

SDVSource Data VerificationSDTMStudy Data Tabulation ModelSOPStandard Operating Procedure

SPC Summary of Products Characteristics

SS Safety Analysis Set

SUSAR Suspected Unexpected Serious Adverse Reaction

Th T helper cell

TNF-α Tumor Necrosis Factor-Alpha

UV-A/B Ultraviolet-A/B

VAS Visual Analogue Scale



Rev: A 

### **Table of Contents**

| 1 | PROTO | COL SUMMARY | 6 |
|----|---------|--------------------------------------------------------|----|
| 2 | STATIS | TICAL METHODOLOGY | 11 |
| 2 | 2.1 Gei | NERAL CONSIDERATIONS | 11 |
| | | BJECT POPULATION | |
| _ | 2.2.1 | Baseline Characteristics/Medical History | |
| | 2.2.2 | Case Disposition | |
| | 2.2.3 | Dose Regimen | |
| | 2.2.4 | Study Populations for Analysis | |
| | 2.2.4.1 | | |
| | 2.2.4.2 | | |
| | 2.2.4.3 | | |
| | 2.2.4.4 | Subgroup Analyses | 13 |
| | 2.2.5 | Study Assessment Time Points | 13 |
| | 2.2.6 | Methods for Handling Missing Data | 14 |
| | 2.2.7 | Safety Monitoring | 15 |
| | 2.2.8 | Statistical Hypotheses | |
| | 2.2.9 | Sample Size Justification | |
| | 2.2.10 | Interim Analyses | |
| | 2.2.11 | Randomization/Unblinding | |
| | 2.2.11. | | |
| | 2.2.11. | | |
| | 2.2.12 | Efficacy Analyses | 16 |
| | 2.2.12. | | |
| | 2.2.12. | = ~~·· | |
| | 2.2.12. | | |
| | 2.2.13 | Safety Analyses | |
| | 2.2.13. | | |
| | 2.2.13. | = | |
| | 2.2.13. | | |
| | | 13.3.1 Serious Adverse Events | |
| | | 13.3.2 Deaths | 23 |
| | 2.2.13. | | 23 |
| | 2.2.13. | | |
| 3 | DOCIN | MENT VERSION CONTROL | |
| - | | | |
| ΑP | PENDIX | A - PROGRAMMING SPECIFICATIONS FOR TABLES AND LISTINGS | 26 |



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

# 1 Protocol Summary

| Title | A Randomised, Double-blind, Placebo-Controlled, Phase 2b Study to Assess the Efficacy and Safety of Orally Administrated DS107 in Patients with Moderate to Severe Atopic Dermatitis. |
|---|---|
| Study Objectives | Efficacy Objective: To compare the efficacy of orally administrated DS107 versus placebo in the treatment of adult patients with moderate to severe Atopic Dermatitis (AD). |
| | Safety Objective: To assess the safety of orally administrated DS107 versus placebo, in adult patients with moderate to severe AD. |
| Primary Endpoint | Proportion of patients achieving an Investigator's Global Assessment (IGA) score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in IGA in treated population compared to placebo population at Week 8. |
| Secondary Endpoint(s) | • Proportion of patients achieving an IGA score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in IGA in treated population compared to placebo population from baseline to Week 2, 4, 6 and 10. |
| | • Proportion of patients achieving a decrease of at least 2 points in IGA in treated population compared to placebo population from baseline to Week 2, 4, 6, 8 and 10. |
| | • Change from baseline in Eczema Area and Severity Index (EASI) in treated population compared to placebo population at Weeks 2, 4, 6, 8 and 10. |
| | • Change from baseline in Numeric Rating Scale (NRS) for Pruritus in treated population compared to placebo population at Weeks 2, 4, 6, 8 and 10. |
| Exploratory Endpoints | • Time to response by Week 8. |
| | • Probability of being in response (PBIR) between Weeks 2 and 8. |
| | Sustained efficacy between Weeks 8 and 10. |
| | • Change from baseline in the Dermatology Life Quality Index (DLQI) score in treated population compared to placebo population at Week 2, 4, 6, 8 and 10 and from Week 8 to Week 10. |



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

| | <ul> <li>Change from baseline in the Patient Orientated Eczema Measure (POEM) score in treated population compared to placebo population at Week 2, 4, 6, 8 and 10 and from Week 8 to Week 10.</li> <li>Change from baseline in the Patient Global Impression of Severity (PGI-S) score in treated population compared to placebo population at Week 2, 4, 6, 8 and 10 and from Week 8 to Week 10.</li> <li>Change from baseline in the Patient Global Impression of Change (PGI-C) score in treated population compared to placebo population at Week 2, 4, 6, 8 and 10 and from Week 8 to Week 10.</li> <li>Plasma DGLA concentrations in treated population compared to placebo population at Baseline/Day 0, Week4, Week 8 and Week 10 (samples to be retained for the potential analysis at a later date).</li> <li>Determination of AD biomarkers in treated population compared to placebo population at Baseline/Day 0 and Week 8/Early</li> </ul> |
|---|---|
| | Termination (samples to be retained for the potential analysis at a later date). |
| Safety Endpoints | <ul> <li>Adverse event (AE) and serious adverse event (SAE) frequency and severity.</li> <li>Safety laboratory parameters (haematology, clinical chemistry).</li> </ul> |
| | Clinical safety examinations (vital signs, physical examination). |
| Test Product, Dose and<br>Mode of Administration | All study medication will be blinded. DS107 capsules will be provided as a capsule containing 500 mg DGLA per unit dose. Placebo will be provided as a matching capsule. This study will involve two dose levels of DS107 for 8 weeks (1g DS107 OD or 2g DS107 OD) and a placebo control (OD) |
| Study Design: | A minimum of 300 patients with moderate to severe AD will be included in this multicenter, double-blind, placebo controlled, 3arm, Phase IIb study. The sample size may be increased at an interim analysis (conducted after n=150 complete Week 8/Exit) to update primary efficacy endpoint assumptions and to achieve at least 80% power and two-sided 5% Type I error. |
| | All patients will sign an informed consent and undergo screening for study eligibility. Patients will be randomized (1:1:1) at baseline visit to either receive 1g DS107 OD once daily or 2g DS107 OD |



Statistical Analysis Plan DS Biopharma DS107G-03

Rev: A 

| | once daily or placeho once daily for & weeks |
|---|---|
| | once daily or placebo once daily for 8 weeks. |
| | Patients will come to the clinic on 7 separate visits: Screening, Baseline (Day0), Week 2, Week 4, Week 6, Week 8 (end of treatment) and Week 10 (follow-up). All patients will exit the study at the Week 10 visit. |
| Inclusion Criteria | 1. Patients with a clinically confirmed diagnosis of active AD |
| | according to Hanifin and Rajka criteria. |
| | 2. Patients with moderate to severe AD at baseline as defined by |
| | an IGA score of minimum 3 at baseline visit. |
| | <ul> <li>3. Patients with an EASI score of ≥12 at screening and baseline.</li> <li>4. Patients with AD covering a minimum 10% of the body surface area at baseline.</li> </ul> |
| | 5. Patients whose pre-study clinical laboratory findings do not |
| | interfere with their participation in the study, in the opinion of the Investigator. |
| | 6. Patients who are able and willing to stop all current treatments |
| | for AD throughout the study (except for allowed emollients). |
| | 7. Patients who are on a stable dose of a bland emollient applied |
| | BD (twice daily) for at least 7 days prior to baseline. |
| | 8. Male or female patients aged 18 years and older on the day of |
| | signing the informed consent form (ICF). |
| | 9. Female patients and male patients with female partners of child bearing potential must use adequate contraception or have a |
| | sterilized partner for the duration of the study. Adequate |
| | contraception is defined as: systemic hormonal contraceptives, |
| | intrauterine device or barrier method of contraception in conjunction with spermicide, or agree to sexual abstinence. |
| | Hormonal contraceptives must be on a stable dose for at least one |
| | month before baseline. |
| | 10. Patients who are able to communicate well with the |
| | Investigator, to understand and comply with the requirements of |
| | the study, and understand and sign the written informed consent. |
| Exclusion Criteria | 1. Patients with other skin conditions that might interfere with AD |
| | diagnosis and/or evaluation (such as psoriasis or current active |
| | viral, bacterial and fungal topical skin infections) as assessed by |
| | the Investigator. |
| | 2. Patients who have used systemic treatments (other than |
| | biologics) that could affect AD less than 4 weeks prior to baseline |
| | visit (Day 0), e.g. retinoids, methotrexate, cyclosporine, |
| | hydroxycarbamide (hydroxyurea), azathioprine and oral/injectable corticosteroids. Intranasal corticosteroids and inhaled |
| | corticosteroids. Intranasal corticosteroids and innated corticosteroids for stable medical conditions are allowed. |
| | cornections for stable medical conditions are allowed. |



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

- 3. Patients who have used any topical medicated treatment for AD two weeks prior to start of treatment/baseline (Day 0) including but not limited to, topical corticosteroids, calcineurin inhibitors, tars, bleach, antimicrobials and bleach baths.
- 4. Patients who use topical products containing urea, ceramides or hyaluronic acid two weeks prior to Day 0.
- 5. Patients who use anti-histamines for AD within 3 days of baseline. Non-sedative anti-histamines for other indications may be used throughout the study provided the patient is on a stable dose for 4 weeks prior to Baseline.
- 6. Patients with the presence of an irregular white cell count as evidenced by eosinophils  $> 0.3 \times 10^9$  /L at the screening visit.
- 7. Patients who have had excessive sun exposure, have used tanning booths or other ultraviolet (UV) light sources four weeks prior to baseline (Day 0) and/or are planning a trip to a sunny climate or to use tanning booths or other UV sources between screening and follow-up visits.
- 8. Patients who have a history of hypersensitivity to any substance in DS107 or placebo capsules.
- 9. Patients who have any clinically significant controlled or uncontrolled medical condition or laboratory abnormality that would, in the opinion of the Investigator, put the patient at undue risk or interfere with interpretation of study results.
- 10. Patients who have a clinically significant impairment of renal or hepatic function.
- 11. Patients with significant uncontrolled cardiovascular, neurologic, malignant, psychiatric, respiratory or hypertensive disease, as well as uncontrolled diabetes and floride arthritis or any other illness that, in the opinion of the Investigator, is likely to interfere with completion of the study.
- 12. Patients with chronic infectious diseases (e.g., hepatitis B, hepatitis C or infection with human immunodeficiency virus).
- 13. Patients with a history of clinically significant drug or alcohol abuse in the opinion of the Investigator in the last year prior to baseline (Day 0).
- 14. Patients who have participated in any other clinical study with an investigational drug within 3 months before the first day of administration of study treatment.
- 15. Patients who have had treatment with biologics as follows: a. Any cell-depleting agents including but not limited to rituximab: within 6 months before the screening visit, or until lymphocyte count returns to normal, whichever is longer, b. Other biologics influencing cell proliferation: within 6 months before the screening



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

| <br>visit. |
|---------------------------------------------------------------------|
| 16. Patients who are pregnant, planning pregnancy, breastfeeding |
| and/or are unwilling to use adequate contraception (as specified in |
| inclusion criterion 7) during the trial. |
| 17. Patients, in the opinion of the Investigator, not suitable to |
| participate in the study. |



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

#### 2 Statistical Methodology

#### 2.1 General Considerations

The objective of this double-blinded Phase 2b study is to assess the efficacy and safety of orally applied DS107 to adults with moderate to severe Atopic Dermatitis. This study uses a randomized (1:1:1, Treatment group A: 1g DS107, Treatment group B: 2g DS107 and Treatment group C: Placebo), double-blind, placebo-controlled parallel group design. Disposition, compliance, demographics, and primary and secondary efficacy results will be presented by treatment group separately for moderate and severe AD as well as for combined groups.

Study medication will be orally applied once daily for 8 weeks. An End of Therapy (EOT) visit will occur at Week 8 for subjects who complete 8 weeks of treatment or earlier if the subject discontinues from the study prematurely. An End of Study (EOS) visit will be conducted at 10 weeks post-treatment for all subjects, even if they withdrew early. For subjects who discontinue early, they will also be asked to return two weeks later for the safety assessments listed at Week 10/Visit 7.

All subjects screened into the study will be assigned a patient identifier number during screening that will be used on all patient documentation. The patient identifier number will contain the site number and the patient number assigned in numerical order at the screening visit (e.g.: 102-10 for the tenth patient screened at the site number 102). Patient numbers will be assigned in ascending order starting with 01. All data will be listed in subject data listings sorted by site and subject number unless otherwise noted. Data tabulations will be prepared as described in the sections below.

All statistical processing will be performed using Statistical Analysis System (SAS®) Version 9.3 or higher, unless otherwise noted. All analyses will be conducted in accordance with ICH E6 and E9 standards and applicable Contract Research Organisation (CRO) Standard Operating Procedures (SOPs). CDISC and SDTM data conventions will be followed; these data sets will include DLQI scoring performed by the data management group and provided to CTDS in the SDTM datasets.

The 2g DS107 treatment group will be tested against the placebo group using a hierarchical approach and if significant at the 0.05 level, then the 1g DS107 treatment group will be tested against the placebo at the 0.05 level, otherwise these will be presented as descriptive statistics.

Baseline values will be defined as the last non-missing measurement prior to dosing with study drug (where baseline record flag='Y' in datasets), unless otherwise specified. Change from baseline will be defined as the post-baseline visit value minus the baseline or previous value unless otherwise specified.



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

#### 2.2 Subject Population

#### 2.2.1 Baseline Characteristics/Medical History

Demographics - gender, age, race (years), ethnicity, country, weight, height, BMI and baseline BSA will be summarized by treatment group for the Full analysis set (FAS) population. Demographics will be displayed separately for the moderate and severe AD as well as overall.

P-values will be provided for the overall global test and each placebo pair (1g DS107 compared to placebo and 2g DS107 compared to placebo) and for comparison of 2g DS107 to 1g DS107. Binary measures (Gender, ethnicity, country and Race—white vs non-white) will be compared using a two-sided Fisher Exact test, while continuous measures (age, weight, height, BMI and baseline BSA) will be compared using ANOVA with Tukey option for the comparison of differences in means between the groups.

Medical History will be tabulated descriptively, including severity of AD, duration of AD (acute, intermediate or chronic) and other relevant medical history. The specific AD medical history reported terms and areas affected will be provided in the listings as text fields.

#### 2.2.2 Case Disposition

All subjects enrolled into the study that are issued a subject number will be accounted for in Subject Disposition. Data will be tabulated by treatment group and the numbers and percentages of subjects in each treatment group who are enrolled, randomized and treated, who comprise the Full Analysis Set (FAS), Safety Analysis Set (SS), and the Per-Protocol Analysis Set (PPS) if there is a >10% loss relative to the FAS analysis populations, and who complete the study or withdraw prematurely along with the reason for discontinuation will be presented. The number of subjects who were seen at each specified study visit will also be tabulated by treatment group and by site. Results will be displayed separately by moderate and severe AD as well as overall.

Protocol deviations (major and minor) will be defined prospectively and will be presented as a listing by treatment group. Major protocol deviations will be tabulated by treatment group.

Reasons for any early withdrawals and the last treatment visit completed prior to discontinuation will be provided in a listing.



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

#### 2.2.3 Dose Regimen

The following three formulations have identical appearance: 1g DS107, 2g DS107 and Placebo in a 1:1:1 ratio, respectively. The medication assigned by randomization will be orally applied by the patients once daily for 8 weeks. Tabulations of exposure to study medication are described in Section 2.2.13.1, Extent of Exposure. Details of study medication use will be provided in a subject data listing.

#### 2.2.4 Study Populations for Analysis

#### 2.2.4.1 Full Analysis Set (FAS)

The FAS consists of all patients who are randomized to the study and received at least one dose of study medication. FAS is the primary analysis population for efficacy endpoints. Analysis will be done according to the treatment patients were randomized to.

#### 2.2.4.2 Safety Analysis Set (SS)

The SS consists of all patients who received at least one dose of the medication. SS is the analysis population for all safety endpoints. Analysis will be done according to the actual treatment patients received.

#### 2.2.4.3 Per-Protocol Analysis Set (PPS)

The PPS is the subset of FAS who completed the study without any major violations. Protocol violations will be assessed for each patient in a blinded fashion prior to database lock at a Blind Data Review Meeting (BDRM), and the PPS will also be finalized during this meeting. PPS is a supportive analysis population for the primary efficacy endpoint. Analysis will be done according to the treatment that patients were randomized to.

#### 2.2.4.4 Subgroup Analyses

Subgroup analyses will be conducted on the primary and secondary endpoints stratifying by severity of atopic dermatitis (moderate or severe), defined as an IGA score of 3=moderate or 4=severe at the Baseline/visit 2 visit, which is consistent with the AD severity used for the entrance criteria in the study. Statistical testing for this subgroup analyses will be limited to the primary efficacy endpoint but summary statistics will be provided for all secondary efficacy endpoints.

#### 2.2.5 Study Assessment Time Points

The study consists of seven protocol-specified visits which will be assessed as nominal visits from an analysis perspective:

# CTDS III

#### FM DM015.1

Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

- Visit 1/Screening visit (Day -30 to -1): Once informed consent has been obtained, the Investigator will assign a Patient Number and the subject will undergo the screening procedures. Following completion of a successful screening visit, patients will begin the comparative treatment period (8 weeks).
- Visit 2/Baseline (Day 0): At the start of the comparative treatment period, after confirmation of continued eligibility, patients will be randomly assigned to one of the three treatment regimens. Study medication is dispensed at Visit 2. The first dose of study medication will be carried out at the site once all baseline assessments have been completed. The patient will carry out their second dose of study medication in the evening of Day 0.
- Visits 3, 4 and 5: Follow-up visits at Week 2 (Day  $14 \pm 2$  days), Week 4 (Day  $28 \pm 2$  days) and Week 6 (Day  $42 \pm 2$  days) respectively.
- Visit 6 End of Treatment (EOT): Week 8 (Day 56 ± 2 days) for subjects who complete 8weeks of treatment; earlier for subjects who discontinue treatment prematurely.
- Visit 7/Week 10: End of Study visit (Day  $70 \pm 3$  days) for all subjects.
- Unscheduled Visits: Unscheduled visits may occur when a patient needs to
  make a visit in between the scheduled visit dates due to an AE, difficulty
  complying with the study protocol requirements, or a significant change in
  their disease state. All procedures that are medically necessary should be
  followed.

# 2.2.6 Methods for Handling Missing Data PROC GENMOD will be used to account for any missing data and early withdrawal for FAS.

The GENMOD procedure will estimate the working correlation from data containing both types of missing values by using the *all available pairs* method, in which all non-missing pairs of data are used in the moment estimators of the working correlation parameters. The resulting covariances and standard errors are valid under the missing completely at random (MCAR) assumption.

A sensitivity analysis will be performed for the Week 8/Exit outcome under the missing at not random (MNAR) assumption for the primary efficacy analyses using the FAS. An extreme analysis will be used to identify the possible outcome considering two scenarios: An extreme analysis will be used to identify the possible outcome considering the worst case for both active treatments and best case for vehicle (Scenario 1) and then the reverse (Scenario 2). If any extreme cases result in statistical significance, then the maximum degree of relaxation per



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

treatment group still reaching statistical significance will be displayed for each scenario. A two-sided Fisher Exact Test will be utilized for these analyses.

#### 2.2.7 Safety Monitoring

No safety monitoring committees are planned for the study.

#### 2.2.8 Statistical Hypotheses

The overall null hypothesis ( $H_0$ ) for each analysis is the equality of the means for the three treatment groups. A global test will be performed across all three treatment groups to allow for a penalty-free comparison of the comparison of the 1g and 2g concentrations against the placebo control. In the event of a global difference (two-sided p<0.05), then the between-treatment comparison of the 2g active treatment group to placebo is performed. If significant (two-sided p<0.05) then the between-treatment comparison of the 1 g active treatment group to the placebo is performed; otherwise the p-values will be regarded as descriptive statistics. The Type I error rate is controlled for by the hierarchical approach. All testing will be two-sided; global tests will be performed at the 0.05 level. Testing between the 2 active groups will be considered descriptive statistics.

#### 2.2.9 Sample Size Justification

The sample size for the topical DS107 Phase IIb study was informed from the post-hoc analysis of the IGA responder data which will be used as the primary endpoint. The positive efficacy data over 4 weeks showed no sign of a plateau and suggests further improvements may be observed at week 8. The sample size was estimated following extrapolation of the IGA responder rate data of the Phase IIa results at weeks 2, 3 and 4 to week 8. Assuming a placebo response rate of 10%, 100 patients per treatment arm (300 patients in total) will be required to detect an absolute difference of 15% in the response rate between an active dose and placebo.

#### 2.2.10 Interim Analyses

An interim analysis is planned to assess primary efficacy endpoint futility and to adjust sample size; EASI will also be evaluated to judge any futility decision. The sample size may be increased at the interim analysis (conducted after n=150 complete Week 8/Exit) to update primary efficacy endpoint assumptions and to achieve at least 80% power and two-sided 5% Type I error.

#### 2.2.11 Randomization/Unblinding

#### 2.2.11.1 Randomization Methodology

At least 300 patients will be randomized to the three blinded treatment groups in a 1:1:1 ratio as follows:

• Treatment group A: 1g DS107 (2 DS107 capsules and 2 placebo capsules) administered once-daily for 8 weeks



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

- Treatment group B: 2g DS107 capsules (4 DS107 capsules) administered once-daily for 8 weeks
- Treatment group C: Placebo capsules (4 placebo capsules) orally administered once-daily for 8 weeks

A randomization list, permuted blocks and stratified by site was generated by HMD Clinical (25 Balmuir Avenue, Bathgate, EH48 4BW, U.K.). The randomization schedule with study drug assignments was generated prior to the start of the study and will be known only to the individuals responsible for labelling the study drug, the statisticians generating the schedule and the IWRS team responsible for implementing the schedule. The IWRS will assign a medication kit number to each patient and the contents will be based on the randomization code.

#### 2.2.11.2 Unblinding

All study site personnel, as well as the personnel involved in the monitoring or conduct of the study, will be blinded to the individual patient treatment assignments. Randomisation details will be kept strictly confidential, accessible only in an emergency to authorized persons, until the time of formal unblinding. The blinded code for the trial will be broken only after all patient data has been recorded and verified and the database locked.

Emergency unblinding will be carried out through the IWRS system with relevant site personnel and pharmacovigilance monitors provided with the required system access to carry out un-blinding.

Any unblinding (and reason for unblinding) prior to database lock will be reported in the final CSR.

#### 2.2.12 Efficacy Analyses

Summary statistics by visit will be provided for all efficacy endpoints. For continuous efficacy endpoints, summary statistics will also be provided for change from baseline at each post-baseline visit. Results for the primary and secondary efficacy endpoints will be presented separately for moderate and severe AD as well as combined across moderate and severe AD strata. Models will include a baseline covariate for moderate/severe for all primary and secondary efficacy analyses. Models will be performed for the primary efficacy endpoint for the separate AD strata but not for the secondary efficacy endpoints.



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

#### 2.2.12.1 Primary Endpoint

The primary efficacy variable will be the proportion of patients achieving an IGA score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in IGA from baseline to week 8. This is a binary endpoint.

The primary endpoint will be analyzed using a Generalised Linear Model (PROC GENMOD) with treatment arm, moderate/severe AD, baseline IGA value, visit and DS treatment dose as factors. The primary analysis will be based on the FAS and repeated for the PPS as a supportive analysis.

This analysis will be performed using SAS PROC GENMOD with code similar to the following:

```
proc genmod data=subjresults descending;
class trt visit subj AD;
model outcome=trt visit trt*visit AD B_IGA /dist=bin;
repeated subject=subj/corr=unstr;
slice trt*visit / sliceby=visit ilink cl diff;
run;
```

where fas= Full Analysis Set (FAS), outcome= patients in each treatment arm at week 8 who achieve an IGA score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in IGA from baseline. B\_IGA is the baseline IGA value. The dist=bin option of the model statement specifies that the logit transformation will be applied to outcome prior to analysis. The cl option specifies that two-sided 95% confidence intervals will be provided and the ilink option specifies the transformation from the logit scale to the probability scale. The between-treatment effects are determined from the diff option of the slice statement. Results will be presented separately for moderate and severe AD for both the FAS and PPS populations. The model will be used to estimate Week 8 effect.

#### 2.2.12.2 Secondary Endpoints

The secondary endpoints are:

• Proportion of patients achieving an IGA score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in IGA in treated population compared to placebo population from baseline to Week 2, 4, 6 and change from baseline to subject's last treatment visit. These analyses will be

# CTDS III

#### FM DM015.1

Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

included in the previous analyses for the primary endpoint for Week 8. A separate model will be performed for the change from baseline to week 10, using the same PROC GENMOD code.

- Proportion of patients achieving a decrease of at least 2 points in IGA in treated population compared to placebo population from baseline to Week 2, 4, 6, 8 and change from baseline to subject's last treatment visit. These analyses will be conducted in the same way as the primary endpoint analysis. A separate model will be performed for the change from baseline to week 10 using the same PROC GENMOD code.
- Change from baseline in Eczema Area and Severity Index (EASI) in treated population compared to placebo population at Weeks 2, 4, 6, 8 and subject's last treatment visit. These will be analyzed using PROC MIXED with treatment arm, moderate/severe AD, baseline IGA value, visit, and DS treatment\*visit as factors. A separate model will be performed for the change from baseline to week 10, using the same PROC MIXED code.

The change from baseline in EASI will be analyzed for the FAS with SAS PROC MIXED using code similar to the following, with CFB\_EASI and B\_EASI representing the change from baseline and the baseline EASI, respectively. Method=ml is the maximum likelihood estimate.

```
proc mixed method =ml data= FAS;
class trt visit subj AD;
model CFB_EASI= trt visit visiti*trt AD B_ EASI /CL;
repeated subject=subj/corr=unstr;
lsmeans trt*visit / diff CL;
run;
```

• Change from baseline in Numeric Rating Scale (NRS) for Pruritus in treated population compared to placebo population at Weeks 2, 4, 6, 8 and subject's last treatment visit. These will be analyzed using PROC MIXED with treatment arm, baseline AD severity, baseline NRS score, visit, and DS treatment\*visit interaction as factors. A separate model will be done for the change from baseline to Week 10, using the same PROC MIXED code.

As NRS is a daily assessment, the analysis of NRS will be performed using the daily average at each visit. At each visit, the average of the NRS values since the previous visit will be computed. Missing values for any

Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

day will be ignored and the between-visit daily average will be computed using non-missing values only. The baseline value will be the average computed during the screening period. This analysis of change from baseline in NRS will be performed the same as the analysis of change from baseline in EASI, with CFB\_NRS and B\_NRS representing the change from baseline in NRS and the baseline NRS, respectively.

#### 2.2.12.3 Exploratory Endpoints

- Time to response by Week 8. A Kaplan-Meier lifetable will be constructed using nominal visits. A Wilcoxon-Gehan test will be used to compare all treatments; p-values will also be computed for each of the three treatment pairs for the primary endpoint using the FAS population. This will be a graph.
- Probability of being in response (PBIR) between Weeks 2 and 8. The PBIR will be computed as a descriptive statistic for the primary endpoint using the FAS population. Each visit will be equally weighted in this analysis. This will be a graph.
- Sustained efficacy between Weeks 8 and 10. This analysis will be endpoint-specific. Binary endpoints will be evaluated using logistic regression (PROC LOGISTIC) controlling for baseline IGA score and baseline AD severity while continuous endpoints will be analyzed using proc GLM controlling for the same factors. A shift table will be created presenting the number and frequencies of subjects in response and the shift from Week 8 to Week 10 for the primary endpoint analysis for both the FAS and PPS populations.
- Change from baseline in the Dermatology Life Quality Index (DLQI) score in treated population compared to placebo population at Week 2, 4, 6, 8 and 10 and from Week 8 to Week 10 and change from baseline to subject's last treatment visit.

DLQI is a set of 10 questions, scored 0=Not at all, 1=A little, 2=A lot, or 3=Very much, or 0=Not relevant, except for Questions 1 and 2 that do not include a response of 'Not Relevant'. Missing responses are assigned '0'. The DLQI total score is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

is impaired. This scoring will be done by the data management group and provided to CTDS in the SDTM datasets.

Mean DLQI will be computed as the Total DLQI divided by the number of questions with non-missing responses. The scoring instructions for DLQI specify that if 2 or more questions are not answered, then the questionnaire will not be scored; this approach is not taken here with Mean DLQI computed instead. Summary statistics for Total DLQI and Mean DLQI will be presented. The analysis of change from baseline in Mean DLQI will be performed the same as the analysis of change from baseline in EASI, with appropriate changes in the variables for change from baseline and Mean DLQI at baseline.

Summary statistics as continuous data and change from baseline will be presented by treatment group and visit for the totals for the 4 sub-scales:

| Symptoms and feelings | Questions 1 and 2 |
|------------------------|-------------------|
| Daily Activities | Questions 3 and 4 |
| Leisure | Questions 5 and 6 |
| Personal relationships | Questions 8 and 9 |

• Change from baseline in the Patient Orientated Eczema Measure (POEM) score in treated population compared to placebo population at Week 2, 4, 6, 8 and 10 and from Week 8 to Week 10 and change from baseline to subject's last treatment visit.

POEM is a set of 7 questions regarding the frequency of conditions related to eczema, with responses of 0 = no days. 1 = 1-2 days, 2 = 3-4 days, 3 = 5-6 days, or 4 = every day. The sum of the scores for the 7 questions is the Total POEM.

Mean POEM is the Total POEM divided by the number of questions with non-missing responses. The scoring instructions for POEM specify that if response to one question is missing, the response for that question will be equated to 0, and if the responses to more than one question are missing, then the questionnaire is not scored; this approach is not taken here with Mean POEM for questions with non-missing responses computed instead. The analysis of change from baseline in Mean POEM will be performed the same as the analysis of change from baseline in EASI, with appropriate changes in the variables for change from baseline and Mean POEM at baseline.

Rev: A 

Summary statistics (counts and frequencies) will be presented by treatment group and visit for categories based on Total POEM of

Clear or almost clear = 0 to 2; Mild eczema = 3 to 7; Moderate eczema = 8 to 16; Severe eczema = 17 to 24; Very severe = 25 to 28.

Shift tables presenting the number and frequency of subjects in each eczema severity category at Week 8 and last treatment visit and Week 8 to Week 10 will be presented by treatment group.

• Change from baseline in the Patient Global Impression of Severity (PGI-S) score in treated population compared to placebo population at Week 2, 4, 6, 8 and 10 and from Week 8 to Week 10 and change from baseline to subject's last treatment visit.

The categories for the PGI-S are: normal, mild, moderate or severe. A Shift table will be created presenting the number and frequencies of subjects in each category and the shift from the follow-up visit to baseline.

Patient Global Impression of Change (PGI-C) is captured at the follow-up visits and is a 7 –point scale assessing the overall status of the patient since the start of the study with responses of 1=very much improved, 2=much improved, 3=minimally improved, 4= no change, 5=minimally worse, 6= much worse and 7=very much worse. Summary statistics (count and frequencies) will be presented by treatment group and visit for the status categories. A shift table presenting the number and frequency of subjects in each category at Week 8 to Week 10 will be presented by treatment group.

• Plasma DGLA concentrations in treated population compared to placebo population at Baseline/Day 0, Week4, Week 8 and Week 10: samples to be retained for the potential analysis at a later date. Details of these analyses will be described in a separate document and the analyses will not be included with the analyses described herein.



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

• Determination of AD biomarkers in treated population compared to placebo population at Baseline/Day 0 and Week8/Early Termination (samples to be retained for the potential analysis at a later date). Details of these analyses will be described in a separate document and the analyses will not be included with the analyses described herein.

#### 2.2.13 Safety Analyses

All subjects enrolled in the study who received at least one dose of the medication will be included in the safety analysis (i.e. Safety Analysis Set).

#### 2.2.13.1 Extent of Exposure

Treatment duration is defined as 8 weeks (Day  $56 \pm 2$  days). The date of the first and last doses of study medication will be collected from information recorded on the study drug admin page of the eCRFs. Study medication is to be orally taken once daily.

Extent of exposure to study medication will be tabulated by treatment group by 2 week intervals. The number of doses of study medication will be summarized by treatment group by each 2 week interval only for those subjects who returned to the clinic for each interval. The expected number of doses per 2 week intervals is 14, based on twice daily dosing. Compliance will be measured by calculating the number of doses/expected number of doses \*100 and presented by treatment group for each interval.

#### 2.2.13.2 Safety Endpoint(s)

The safety objective is to compare the safety of orally administered DS107 capsules (1g & 2g) versus placebo, in the treatment of adult patients with moderate to severe AD. Results will be pooled for 1g and 2g treatment groups as well.

#### 2.2.13.3 Adverse Events

Counts and percentages of subjects who experienced any of the following will be presented by treatment group, as well as a total DS107 treatment group that includes both the 1g and 2g DS107 subjects: any AE, any IMP related AE, any AE requiring modification of study medication dosing (dose reduced, drug interrupted), discontinuations of study participation due to an AE (drug withdrawn), any serious adverse events (SAE), deaths, or IMP related SAEs. Only those adverse events determined to be treatment emergent (TEAE) will be presented (where Qlabel="Treatment").



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

Emergent" from the SUPPAE SDTM dataset). Treatment emergent adverse events are those events with the date of AE onset being greater than or equal to the date of the first dose date of study drug. A two-sided Fisher Exact test will be utilized for an overall global test and for the pairwise comparisons of each treatment compared to placebo.

Verbatim terms on the case report forms will be coded to preferred term (PT) and related system organ class (SOC) using MedDRA Coding Dictionary Version 19.1. The number and percentage of subjects who experience treatment-emergent adverse events (TEAE) will be tabulated by System Organ Class (SOC) and Preferred Term (PT) within each treatment group. The number of events will be tabulated by System Organ Class (SOC) and Preferred Term (PT) within each treatment group. In addition, a tabulation of adverse events that occur at a frequency of 2% or greater at the SOC or PT level will be prepared. A two-sided Fisher Exact test will be performed on system organ class (SOC) with a 2% or greater frequency to facilitate evaluation of potential safety differences among treatments.

Adverse events will be counted only once for a subject within each Preferred Term and System Organ Class; thus, since a subject may have more than one Preferred Term within an SOC, percentages of PT may not sum to the percentage in the SOC. If a subject reports a Preferred Term multiple times with differing severities (mild, moderate or severe), only the most severe is counted but all events will be counted. If a subject reports a Preferred Term multiple times with differing relationships to IMP, only the one that is related to IMP is counted.

#### 2.2.13.3.1 Serious Adverse Events

The number and percentage of subjects experiencing a Serious Adverse Event (SAE) will be tabulated by SOC and PT within each treatment group and overall. SAEs will be counted only once for a subject within each PT and SOC.

#### 2.2.13.3.2 Deaths

A listing of subjects who die while on study will be prepared along with the adverse event associated with the cause of death.

# 2.2.13.3.3 Interruptions or Discontinuations of Study Medication Due to an AE

A listing of subjects who have changes to their study medication dosing (dose reduced, interruptions or discontinuations) will be prepared.

Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

#### 2.2.13.4 Laboratory Data

Any laboratory test results considered to be clinically significant by the Investigator will be captured as an adverse event. All clinical laboratory values (haematology and biochemistry) will not be tabulated but will be listed for each patient by treatment group and visit. Values outside the laboratory normal ranges will be listed separately by patient and treatment group with associated comments as to their clinical significance.

# 2.2.13.5 Vital Signs, Physical Findings, and Other Observations Related to Safety

Vital signs are collected at the screening, visit 2/baseline and the follow-up visits. Temperature (°C), systolic and diastolic blood pressure (mmHg) and heart rate (BPM) will be tabulated by treatment group using the baseline value (where baseline record flag= 'Y') and end of study (week 10). Change from end of study to baseline will be presented as descriptive statistics.

Physical Examination Findings will be presented in the listings but not tabulated.

Concomitant Medications will be coded per the WHO Drug dictionary (version effective March 2017 and provided to CTDS in the SDTM CM dataset. Concomitant Medications will be tabulated by treatment group, Drug Class (pharmacological level, ATC3) and Drug Name (chemical substance level, ATC5). These data will be provided in subject data listings along with the verbatim drug term and usage details.



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

### **3 Document Version Control**

# **Revision History:**

| REVISION | RELEASE | AUTHOR | SUMMARY OF CHANGES |
|----------|-----------|---------------|--------------------|
| | DATE | | |
| A | 17Jul2017 | CTDS/P. Lavin | Initial Version |



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

#### **Appendix A - Programming Specifications for Tables and Listings**

The following specifications will be used in the production of tables and listings.

#### 1. Page Setup

Unless otherwise noted, tables and listings will use landscape orientation. Margins will be at least 1.5 inches on the bound side and at least 1 inch on the other three sides.

The following header information should be included:

- Upper left: Sponsor name and protocol number
- Center: CONFIDENTIAL
- Upper right: Page number shown as Page n of N. Page numbers should be sequential within a table or listing.

#### The footer should include:

- The name of the SAS program used to generate the output along with the run date/time and the words "by CTDS".
- For tables, the corresponding listing number(s).

#### 2. Footnotes

Unless otherwise specified, footnotes should appear on all pages within the table.

#### 3. Font

Font will be 8-point Arial, or smaller if needed for space constraints. If possible, small tables should appear on one page. If tables continue on to multiple pages, there should be a page break after an assessment so that all the statistics for an assessment appear on the same page.

#### 4. Tables

Table titles should reflect the content of the table. Under the main title, in parentheses, the name of the analysis population being summarized should appear.

#### 4.1 Summary Statistics - Continuous Data

Unless otherwise noted, the mean and median and confidence interval (CI) of a set of values should be printed out to one decimal place more than the original value. The standard deviation should be printed out to 2 decimal places more than the original value. The number of subjects on whom the parameter is assessed should appear. Minimum and maximum should be consistent with the original value. P-values will be expressed as 4 decimal places. Any p-values that get calculated as 0.0000 should be expressed as p-value <0.0001.

#### 4.2 Summary Statistics - Categorical Data



Statistical Analysis Plan DS Biopharma DS107G-03 Rev: A 

Numbers of subjects are reported as whole numbers. Null counts are represented as 0. Table percentages should be reported to one decimal unless otherwise noted. Null percentages should be reported as 0.0%.

For all categories, the total number of subjects with data will be presented as N and the number of subjects with non-missing data will be used as the denominator for the calculation of the percentages, unless otherwise noted.

#### 5. Subjects Included in Listings

In general, subject data listings should include all subjects who signed the informed consent. If a listing includes a subset of subjects who meet a certain condition (eg, subjects with SAEs) then this should be clear from the title of the listing. If there are no subjects who meet the condition (eg, no subjects with SAEs) for either the tables or the listings, then a page marker should appear stating that no subjects met the criteria.